CLINICAL TRIAL: NCT02216617
Title: A Phase I Study Evaluating the Combination Afatinib With Docetaxel and Cisplatin (TPA) in Induction Chemotherapy in Locally Advanced Squamous Cell Carcinoma of the Upper Aerodigestive Tract
Brief Title: Evaluation of the Tolerance of Afatinib in Combination With Docetaxel and Cisplatin in LAHNSCC Induction Chemotherapy
Acronym: TAPIS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Groupe Oncologie Radiotherapie Tete et Cou (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GORTEC 2013-01; 2013-002876-42 (EudraCT Number)
Record Dates: First submitted 2014-08-07; First posted 2014-08-15 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: HNSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Docetaxel; Cisplatin; Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Induction chemotherapy TPA (Experimental): 3 Cycles of induction chemotherapy TPA : (Taxotere, Cisplatin, Afatinib)
  1 cycle = 3 weeks, three cycles of treatment in total (or 9 weeks)
  Docetaxel 75 mg / m2 at D1 Cisplatin 75 mg / m 2 at D1 Afatinib: x mg / day D2 to D21 by level: (Level 1: 20 mg / day; Level 2: 30 mg / day; Level 3: 40 mg / day)
  Interventions: Drug: Taxotere, Cisplatin, Afatinib

INTERVENTIONS:
Drug: Taxotere, Cisplatin, Afatinib

SUMMARY:
The purpose of the study is to determine the maximum tolerated dose (MTD) of afatinib administrated in combination with docetaxel (Taxotere®) and cisplatin in induction chemotherapy of locally advanced head and neck carcinoma in order to move to a phase II, allowing the comparison with standard induction chemotherapy TPF.

It is a multicentric, national, opened, not-randomized phase Ib. Three doses of afatinib (20, 30 and 40 Mg per day) will be studied in combination with the fixed standard doses of docetaxel and cisplatin. For each dose level, beginning with smallest (20 Mg per day of afatinib), 3 to 6 patients will be treated at maximum, i.e. 3 cycles of three weeks treatment each one (9 weeks on the whole). The next dose level will be studied only if the previous dose is well tolerated for the period of the first 4 weeks observation of the treatment (1st cycle more first week of the 2nd cycle). Once the MTD is determined, four additional patients will be treated with this dose. A maximum of 22 patients should be included in this study. The total duration of the study is estimated at 18 months. In case of major safety problems, the study may be stopped earlier. In short, the preclinical data, pharmacological and clinical on afatinib indicate that the benefit-risk ratio can be regarded as positive and that the association of afatinib with cisplatin and docetaxel could be effective in patients with head and neck squamous cell carcinoma potentially resulting in an extension of time to progression.

DETAILED DESCRIPTION:
Cancers of the upper aerodigestive tract correspond in the Western countries about 5% of cancers. They are treated by surgery, radiotherapy, and chemotherapy. Although progress in radio chemotherapy have reduced mortality and increase the rates of organ preservation in patients with locally advanced head and neck cancers, they have metastatic risk or particularly high local recurrence. The induction chemotherapy is a first-line treatment of cancer in which the patient receives doses of chemotherapy allowing to obtain a significant reduction in tumor size, and thus to avoid the surgery and to treat the tumor then by radiotherapy alone or combine by certain drugs. The standard treatment of induction chemotherapy currently used for the carcinoma of aerodigestive tract is TPF compose of 3 drugs: the docetaxel (or Taxotere®, T), the cisplatin (P) and the 5-fluorouracil (or 5FU, F). Despite of the relative efficacy of this treatment, which provides a survival benefit, it is necessary to find a combination of induction to be more effective and less toxic. That is why this study intended to check if a new combination called TPA in which the fluorouracil (F) is replaced by the afatinib (A), will be more beneficial. The afatinib is a powerful and irreversible inhibitor of the EGFR (human Epidermal Growth Factor Receptor type 1), HER2 and HER 4. The EGFR is associated with a pejorative prognosis and resistance to the treatments through its role in the proliferation (multiplication of tumoral cells), the cell survival and replication and angiogenesis (process of growth of new blood-vessels, vital in the growth of the malignant tumors). Afatinib has proved effective in patients in with local recurrence or metastatic squamous cell carcinoma of the head and neck after first line cisplatin based and tolerance is correct.

The rational of this study is based on the following elements:

* Cisplatin and docetaxel on the one hand and the afatinib on the other hand have proved effectiveness in head and neck cancers. The tolerance of their association is not known.
* In addition, several broad randomized trials have shown that it is possible to improve the effectiveness of induction chemotherapy in locally advanced head and neck carcinoma by the addition of Taxotere® to the cisplatin-5FU.
* Independently, it has been shown in carcinoma of the upper aerodigestive tract with recurrence or metastatic, that an anti-EGFR targeted therapy by cetuximab could improve the effectiveness of chemotherapy with cisplatin-5FU More recently, Taxotere® and Cisplatin + Cetuximab (or Erbitux®) combination for the treatment of head and neck squamous cell carcinoma has been tested in a broad study of phase II showing the good feasibility of this combination and a particularly high rate of tumoral response.
* Finally a comparative study of cetuximab versus afatinib showed an advantage in terms of tumoral response in support of afatinib.

From all these observations, the investigators can hypothesize that the addition of afatinib to the docetaxel and the cisplatin could be an induction treatment for locally advanced carcinoma both innovating and promising. Indeed, this regimen appears optimized in terms of efficiency, incorporating both the combination of the most active cytotoxic agents, Taxotere® and the cisplatin, but also potentially more effective than Erbitux®.

The purpose of the study is to determine the Maximum Tolerated Dose (MTD) of afatinib administrated in combination with docetaxel (Taxotere®) and cisplatin in induction chemotherapy of locally advanced head and neck carcinoma in order to move to a phase II, allowing the comparison with standard induction chemotherapy TPF.

It is a multicentric, national, opened, not-randomized phase Ib. Three doses of the afatinib (20, 30 and 40 Mg per day) will be studied in combination with the fixed standard doses of the docetaxel and the cisplatin. For each dose level, beginning with smallest (20 Mg per day of afatinib), 3 to 6 patients will be treated at maximum, i.e. 3 cycles of three weeks treatment each one (9 weeks on the whole). The next dose level will be studied only if the previous dose is well tolerated for the period of the first 4 weeks observation of the treatment (1st cycle and first week of the 2nd cycle). Once the MTD is determine, four additional patients will be treated with this dose. A maximum of 22 patients should be included in this study. The total duration of the study is estimated at 18 months. In case of major safety problems, the study may be stopped earlier. In short, the preclinical data, pharmacological and clinical on afatinib indicate that the benefit-risk ratio can be regarded as positive and that the association of afatinib with cisplatin and docetaxel could be effective in patients with head and neck squamous cell carcinoma potentially resulting in an extension of time to progression.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤70 years
* Patient in first line treatment of Locally Advanced HNSCC, histologically proven non-metastatic
* At least one measurable lesion (RECIST)
* Eligible patient for standard induction chemotherapy in the opinion of the investigator; PS ECOG < 2

Adequacy functioning of organs, including:

* Left ventricular function with ejection fraction at rest > 50% or as normal institutional values Haematological function
* Absolute neutrophil count (ANC) >1,500/mm3 Special cases: ANC> 1,000/mm3 in the opinion of the investigator and discussion with the sponsor; Platelets ≥ 75,000/mm3; Hemoglobin> 10g/dl

Liver function:

•Total bilirubin ≤ 1.5 x ULN; patients with Gilbert's syndrome must have a total bilirubin <4 x ULN; SGOT and SGPT ≤ 3 x ULN or SGOT and SGPT ≤ 5 x ULN in case liver abnormalities; Alkaline phosphatase <2.5 x ULN

Kidney function:

•Serum creatinine <110 umol/L or creatinine clearance > 45 ml/min (Cockcroft method)

General:

* Men and women of childbearing potential must agree to use a reliable contraception throughout treatment and at least 6 months after the end of treatment. Women in peri-menopause should be least 24 months of amenorrhea.
* Ability to take oral medication in the opinion of the investigator; Patient affiliated to a social security system; signed informed consent form.

Exclusion Criteria:

•Previous treatment with chemotherapy, radiation therapy or targeted therapy for head and neck cancer; uncontrolled Respiratory, cardiac, hepatic or renal diseases.

Significant cardiovascular disease like:

* Cardiovascular Abnormalities considered clinically important as congestive heart failure NYHA stage ≥ III, unstable angina or myocardial infarction within the past 6 months, or arrhythmia low controlled, uncontrolled hypertension by treatment (systolic BP ≥ 160 mmHg and/or diastolic BP≥ 90 mmHg).
* Impairment of left ventricular function with an ejection fraction ≤ 50%; Stroke within 6 months prior to inclusion.
* Severe thromboembolic history within 6 months prior to inclusion.
* Lengthening of the corrected QT interval with QTc> 480 msec according to the formula Bazet; Bradycardia; Electrolyte disturbances

Respiratory disease of type:

•interstitial lung disease; Pulmonary fibrosis

Viral disease of type:

•Active infection or hepatic B virus or hepatitis C known carrier of HIV.

Recent digestive disorder with diarrhea such as:

* Any history or presence of gastrointestinal disorders with uncontrolled diarrhea as a major symptom that may affect the absorption of drug tested in the opinion of the investigator (eg disease Crohn's disease, diarrhea CTCAE grade ≥ 2)
* Any past or present condition that would compromise the patient's ability to comply with the study or which would interfere with the evaluation of the effectiveness and the safety of the study.
* Other severe disease or condition associated with non-oncological origin likely to be incompatible with the protocol in the judgment of the investigator.
* Patient already included in another clinical trial with an experimental molecule; Persons deprived of liberty or under guardianship or as backup justice.
* Patient requiring prohibited concomitant treatments with study.
* Any cons-indication to treatment with Taxotere or Afatinib or cisplatin.
* Known hypersensitivity to Afatinib or excipients the study drugs; Major surgery within 4 weeks before taking treatment; Use of products in a clinical study during the 4 weeks preceding inclusion.

Radiation therapy within 4 weeks before inclusion.

•Presence and / or history (in the past 3 years) cancer except Basal cell skin cancer, cervical carcinoma in situ and prostate cancer in situ; Pregnant or during breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-08-06; Primary Completion 2015-07 (Actual); Study Completion 2015-09-15 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | During the first 4 weeks of treatment for each patient of the bearing.
  The main objective is to determine the Maximum Tolerated Dose (MTD) of afatinib in combination with docetaxel and cisplatin chemotherapy TPA induction in locally advanced head and neck carcinomas in order to move a phase II for comparison with induction chemotherapy "of reference "TPF (Taxotere, cisplatin and 5-fluorouracil).

SECONDARY OUTCOMES:
Tolerance | 12 weeks
  Tolerance: Toxicity will be evaluated by NCI CTCAE V4.03. scale
Efficacy | 12 weeks
  Efficacy: Objective tumor response will be evaluated through RECIST V1.1

OTHER OUTCOMES:
Correlation between nutritional status and toxicity | 12 weeks
  Objective is to correlate the values of body fat / lean mass determined by CT-scan to the nutritional status of the patients and toxicities.

CONTACTS AND LOCATIONS:
Overall Officials: Didier CUPISSOL, MD, Study Chair — GORTEC
Locations (1):
- ICM Val d'Aurelle, Montpellier, Montpellier, France

REFERENCES:
- See also: Related Info — http://www.gortec.fr/